CLINICAL TRIAL: NCT01469767
Title: Efficacy of Fluocinonide Cream 0.1% (Vanos(R)) in Reducing Itch in Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: Medicis Pharmaceutical Corporation (Industry)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00018876
Record Dates: First submitted 2011-11-07; First posted 2011-11-10 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-08

CONDITIONS: Atopic Dermatitis
Keywords: eczema; itch; scratching; actigraphy; adherence
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Pruritus | interventions — Fluocinonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fluocinonide cream (Experimental): Subjects will apply fluocinonide cream 0.1% twice daily for 5 days.
  Interventions: Drug: Fluocinonide cream

INTERVENTIONS:
Drug: Fluocinonide cream — Fluocinonide cream 0.1% applied twice daily for 5 days.
  Other Names: Vanos

SUMMARY:
The purpose of this study is to assess the efficacy of short-term treatment with fluocinonide cream 0.1% (Vanos®) in the treatment of atopic dermatitis (AD).

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy of short-term treatment with fluocinonide cream 0.1% (Vanos®) in the treatment of atopic dermatitis (AD). Our hypothesis is that subjects will have a reduction in Investigator's Global Assessment scores at Day 7 and Day 14 compared to Baseline.

Secondary objectives include the use of actigraphy monitoring to determine the ability of Vanos® cream to reduce itch, and thus nocturnal scratching, in AD. Our hypothesis is that subjects will have a reduction in nocturnal scratching activity, as measured by actigraphy movement count per hour, at Day 7 and Day 14 compared to Baseline. Other secondary outcome measures include Eczema Area and Severity Index (EASI) score, body surface area involvement and Visual Analog Scale for itch. The investigators hypothesize that each of these measures will be improved at Day 7 and Day 14 compared to Baseline.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with mild to severe atopic dermatitis, 12 years of age or older, that agree to participate and provide written consent (parent permission and assent if applicable).
* Have an Investigator Global Assessment of mild to severe atopic dermatitis (IGA rating of 2 through 4 in the Investigator Global Assessment).
* Visual Analog Scale of Itch score at Baseline must be greater than or equal to 50 on a 100-point scale.
* Percentage of overall body surface area of involvement (BSA) must be ≥2%.
* Women of childbearing potential will be allowed to participate in the study, and will be required to use at least one form of birth control.

Exclusion Criteria:

* Use within four weeks from Baseline any systemic anti-inflammatory medication, which may influence study outcome, such as systemic corticosteroids.
* Application or use within two weeks of Baseline topical corticosteroid medications or topical anti-inflammatory medication, which may influence study outcome.
* Presence of a concurrent medical condition, which is determined by the investigator to potentially interfere with study outcomes or patient assessments.
* Introduction of any other prescription medication, topical or systemic, for atopic dermatitis while participating in the study.
* Use of anti-histamines while participating in the study will not be permitted unless the subject meets criteria for anti-histamine use on the VAS scale. Additionally, the subject must remain on a stable dose of anti-histamine throughout the study period. If a patient meets such criteria for anti-histamine use, this will be noted in the subject's chart.
* Amount of disease involvement that would require >60 gm of cream in a 1 week period.
* Subjects with known allergy or sensitivity to topical Vanos® cream or components.
* Pregnant women
* Women who are breastfeeding

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2013-08-17 (Actual); Study Completion 2013-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluocinonide Cream
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fluocinonide Cream
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 6
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: IGA
Description: Investigator's Global Assessment of atopic dermatitis integrates all lesions for overall score. This measure is commonly used to quantify disease severity and most resembles assessments performed in the clinic setting. Score ranges from '0' = Clear to '5' = Very Severe Disease
Time Frame: 14 days
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Fluocinonide Cream
Number analyzed (Participants) | 10
units on a scale | 1 [1 to 3]

2. Secondary Outcome: Actigraphy
Description: Actigraphy Movement Count per Hour:Subjects will be asked to wear an actigraphy monitor on each wrist for the duration of the 14-day study. These monitors appear and function similarly to a wristwatch. The actigraph provides a continuous measure of wrist activity and may be used to quantify nocturnal scratching behavior. A piezoelectric accelerometer records the integration of intensity, amount, and duration of stimuli in all 3 dimensions of wrist movement. Measurements are taken at 32 Hz and a summation value is recorded at the end of each 30-second epoch. The number of 30-second epochs with movement (in which acceleration was detected irrespective of the magnitude of the acceleration) is recorded and summed to give a movement score. This is divided by the duration of time in bed to produce a movement count per hour, which is a sensitive quantitative measure of scratch-associated activity.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: Movement count per hour
Arm/Group | Fluocinonide Cream
Number analyzed (Participants) | 10
Movement count per hour | 85.7 (3.2)

3. Secondary Outcome: EASI
Description: Eczema Area and Severity Index Score:Disease severity will be assessed with the Eczema Area and Severity Index (EASI).This measure is commonly used and well validated instrument of eczema severity. It is weighted for area in each of the four body regions and scores erythema, excoriation, induration/papulation, and lichenification. The total are summed for one total EASI score. .The total scores range from 0 (no Eczema) -72 (most severe Eczema)."
Time Frame: 14 days
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Fluocinonide Cream
Number analyzed (Participants) | 10
units on a scale | 2.2 [0.2 to 23.2]

4. Secondary Outcome: BSA
Description: Body Surface Area of atopic dermatitis. The BSA is measured as the total percent of the entire body with atopic dermatitis involved, so the scores range from 0% to 100% of total body involvement.
Time Frame: 14 days
Measure: Mean (Full Range); unit: Percent BSA
Arm/Group | Fluocinonide Cream
Number analyzed (Participants) | 10
Percent BSA | 5.5 [1 to 55]

5. Secondary Outcome: VAS
Description: Visual Analog Scale for itch: A 100 millimeter (mm) Visual Analog Scale (VAS) will be used to measure itch intensity. VAS is a self-report tool that is designed to present to the respondent a rating scale with minimum constraints. VAS data is recorded as the number of mm from the left of the line with the range 0-100 mm. The Visual Analog Scale is anchored with the verbal descriptions of "no itch" on the left and "the most intense itch imaginable" on the right.
Time Frame: 14 days
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Fluocinonide Cream
Number analyzed (Participants) | 10
units on a scale | 41 [0 to 100]

ADVERSE EVENTS:
Arm/Group | Fluocinonide Cream
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes